CLINICAL TRIAL: NCT05831631
Title: Immunophenotype Characterization of Circulating and Tumor Infiltrating Immune Cells in Malignant Brain Tumors.
Brief Title: Characterization of Circulating and Tumor-infiltrating Immune Cells in Malignant Brain Tumors
Status: Recruiting | Type: Observational
Sponsor: Pietro Mortini, MD, Prof. (Other)
Responsible Party: Sponsor-Investigator, Pietro Mortini, MD, Prof., Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: NCH 02-2022
Record Dates: First submitted 2023-03-16; First posted 2023-04-26 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Brain Tumor, Primary; Brain Tumor - Metastatic
Keywords: Immunophenotype; Primary and secondary brain tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for lymphocyte extraction and immunophenotype detection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Included patients: The study population will comprise 200 (two hundred) adult patients candidate to neurosurgical treatment for newly diagnosed malignant brain tumors, able to express an informed consent.
  Interventions: Diagnostic Test: Circulating leukocytes immunophenotype; Diagnostic Test: Tumor sampling

INTERVENTIONS:
Diagnostic Test: Circulating leukocytes immunophenotype — Blood samples will be tested with flow cytometry in order to characterize leukocyte subpopulations and to evaluate the circulating immunophenotype
Diagnostic Test: Tumor sampling — Immunohistochemical analysis will be performed on tumor samples in order to characterize immune T cells distribution within the tumor.

SUMMARY:
The goal of this observational study is to characterize the circulating leukocyte profile and the immune T cells distribution within the tumor in patients with malignant brain tumors and to correlate these findings with the oncological outcome.

Participants will be subjected to blood sampling before surgery and for 12 months of follow-up. Additional sampling and analysis will be performed on tumor samples.

DETAILED DESCRIPTION:
High-grade gliomas are the most frequent type of primary brain tumor in adults, and among them, glioblastoma multiforme (GBM) is the most malignant with an associated poor prognosis. Although significant advances have been achieved in GBM biology comprehension, patients' life expectancy is still limited to 18 months.

Brain metastases (BM) are the most frequent neoplasm in the CNS; it is estimated that up to 14% of all newly diagnosed cancers will soon or later metastasize into the brain.

A variety of mechanisms to escape a tumor-specific T cell-mediated immune response have been identified in glioma and other cancer entities.

This project is an observational, prospective, monocentric study on patients candidates for neurosurgical procedures for brain malignant tumors with additional collection of biological material. With the present study, we aim to characterize the phenotype of both circulating- and tumor-infiltrating- immune cells at the diagnosis and their changes during disease progression and after treatment in primary and secondary brain tumors.

Samples will be taken at baseline (before surgery) and at time-points: 3, 6, 9, 12 months

ELIGIBILITY:
Inclusion criteria:

* Adult patients (≥18 years)
* Able to express informed consent
* With primary or secondary malignant brain tumor
* Requiring neurosurgical treatment (radiosurgery, stereotactic biopsy, surgery)

Exclusion Criteria:

* Patients who do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of malignant brain tumor (primary or secondary) and meeting the criteria for undergoing neurosurgical treatment (radiosurgery, stereotactic biopsy, surgery).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Baseline leucocytes count | Baseline
  Leucocytes count (10^3/ml), total lymphocytes count (10^3/ml)
Baseline leucocytes immunophenotype | Baseline
  Determination of different leucocyte subpopulations (%)
Baseline tumor-infiltrating lymphocytes count | After surgery (tumor sampling)
  Infiltrating lymphocytes count (10^3/ml)
Baseline tumor-infiltrating leucocytes immunophenotype | After surgery (tumor sampling)
  Infiltrating T-cell subpopulations (%)

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Mortini, MD, Prof., Study Director — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olar A, Aldape KD. Using the molecular classification of glioblastoma to inform personalized treatment. J Pathol. 2014 Jan;232(2):165-77. doi: 10.1002/path.4282. PMID 24114756
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Wang W, Shi G, Ma B, Hao X, Dong X, Zhang B. Chemotherapy for Adults with Malignant Glioma: A Systematic Review and Network Meta-Analysis. Turk Neurosurg. 2017;27(2):174-181. doi: 10.5137/1019-5149.JTN.15462-15.0. PMID 27337236
- [Background] Barnholtz-Sloan JS, Sloan AE, Davis FG, Vigneau FD, Lai P, Sawaya RE. Incidence proportions of brain metastases in patients diagnosed (1973 to 2001) in the Metropolitan Detroit Cancer Surveillance System. J Clin Oncol. 2004 Jul 15;22(14):2865-72. doi: 10.1200/JCO.2004.12.149. PMID 15254054
- [Background] Lowery FJ, Yu D. Brain metastasis: Unique challenges and open opportunities. Biochim Biophys Acta Rev Cancer. 2017 Jan;1867(1):49-57. doi: 10.1016/j.bbcan.2016.12.001. Epub 2016 Dec 6. PMID 27939792
- [Background] Kromer C, Xu J, Ostrom QT, Gittleman H, Kruchko C, Sawaya R, Barnholtz-Sloan JS. Estimating the annual frequency of synchronous brain metastasis in the United States 2010-2013: a population-based study. J Neurooncol. 2017 Aug;134(1):55-64. doi: 10.1007/s11060-017-2516-7. Epub 2017 May 31. PMID 28567587
- [Background] Kim YH, Jung TY, Jung S, Jang WY, Moon KS, Kim IY, Lee MC, Lee JJ. Tumour-infiltrating T-cell subpopulations in glioblastomas. Br J Neurosurg. 2012 Feb;26(1):21-7. doi: 10.3109/02688697.2011.584986. Epub 2011 Jun 27. PMID 21707245
- [Background] Lohr J, Ratliff T, Huppertz A, Ge Y, Dictus C, Ahmadi R, Grau S, Hiraoka N, Eckstein V, Ecker RC, Korff T, von Deimling A, Unterberg A, Beckhove P, Herold-Mende C. Effector T-cell infiltration positively impacts survival of glioblastoma patients and is impaired by tumor-derived TGF-beta. Clin Cancer Res. 2011 Jul 1;17(13):4296-308. doi: 10.1158/1078-0432.CCR-10-2557. Epub 2011 Apr 8. PMID 21478334
- [Background] Kmiecik J, Poli A, Brons NH, Waha A, Eide GE, Enger PO, Zimmer J, Chekenya M. Elevated CD3+ and CD8+ tumor-infiltrating immune cells correlate with prolonged survival in glioblastoma patients despite integrated immunosuppressive mechanisms in the tumor microenvironment and at the systemic level. J Neuroimmunol. 2013 Nov 15;264(1-2):71-83. doi: 10.1016/j.jneuroim.2013.08.013. Epub 2013 Aug 31. PMID 24045166
- [Background] Sayour EJ, McLendon P, McLendon R, De Leon G, Reynolds R, Kresak J, Sampson JH, Mitchell DA. Increased proportion of FoxP3+ regulatory T cells in tumor infiltrating lymphocytes is associated with tumor recurrence and reduced survival in patients with glioblastoma. Cancer Immunol Immunother. 2015 Apr;64(4):419-27. doi: 10.1007/s00262-014-1651-7. Epub 2015 Jan 3. PMID 25555571
- [Background] Mauldin IS, Jo J, Wages NA, Yogendran LV, Mahmutovic A, Young SJ, Lopes MB, Slingluff CL Jr, Erickson LD, Fadul CE. Proliferating CD8+ T Cell Infiltrates Are Associated with Improved Survival in Glioblastoma. Cells. 2021 Dec 1;10(12):3378. doi: 10.3390/cells10123378. PMID 34943886
- [Background] Vilarino N, Bruna J, Bosch-Barrera J, Valiente M, Nadal E. Immunotherapy in NSCLC patients with brain metastases. Understanding brain tumor microenvironment and dissecting outcomes from immune checkpoint blockade in the clinic. Cancer Treat Rev. 2020 Sep;89:102067. doi: 10.1016/j.ctrv.2020.102067. Epub 2020 Jul 7. PMID 32682248
- [Background] Mohme M, Schliffke S, Maire CL, Runger A, Glau L, Mende KC, Matschke J, Gehbauer C, Akyuz N, Zapf S, Holz M, Schaper M, Martens T, Schmidt NO, Peine S, Westphal M, Binder M, Tolosa E, Lamszus K. Immunophenotyping of Newly Diagnosed and Recurrent Glioblastoma Defines Distinct Immune Exhaustion Profiles in Peripheral and Tumor-infiltrating Lymphocytes. Clin Cancer Res. 2018 Sep 1;24(17):4187-4200. doi: 10.1158/1078-0432.CCR-17-2617. Epub 2018 Feb 14. PMID 29444930
- [Background] Gagliardi F, De Domenico P, Snider S, Roncelli F, Pompeo E, Barzaghi LR, Bulotta A, Gregorc V, Lazzari C, Cascinu S, Finocchiaro G, Mortini P. Role of stereotactic radiosurgery for the treatment of brain metastasis in the era of immunotherapy: A systematic review on current evidences and predicting factors. Crit Rev Oncol Hematol. 2021 Sep;165:103431. doi: 10.1016/j.critrevonc.2021.103431. Epub 2021 Jul 27. PMID 34324961